CLINICAL TRIAL: NCT02909413
Title: Comparison of Desflurane With Sevoflurane for School-age Children in Postoperative Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yingjie Du, Anesthesiology residency, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: DES VS. SEV
Record Dates: First submitted 2016-04-27; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: desflurane; sevoflurane
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Desflurane (Experimental): Anesthesia maintenance: After endotracheal intubation, patients will be randomized into Desﬂurane for maintenance. The gas flow rate of Desflurane group is 2 L/min, include 50％ O2 and 4～5％ Desflurane.
  Interventions: Drug: Desﬂurane
- Group Sevoflurane (Active Comparator): Anesthesia maintenance: After endotracheal intubation, patients will be randomized into sevoﬂurane for maintenance. The gas flow rate of Sevoflurane group is 2L/ min, include 50％O2 and 1.7-2.0% Sevoflurane.
  Interventions: Drug: sevoﬂurane

INTERVENTIONS:
Drug: Desﬂurane — Anesthesia maintenance: After endotracheal intubation, half of the patients will be randomized into Desﬂurane Group. The gas flow rate of Desflurane group is 2 L/min, include 50％ O2 and 4～5％ Desflurane.
  Arms: Group Desflurane
Drug: sevoﬂurane — Anesthesia maintenance: After endotracheal intubation, half of the patients will be randomized into Sevoﬂurane Group. The gas flow rate of Desflurane group is 2 L/min, 50％O2 and 1.7-2.0% Sevoflurane.
  Arms: Group Sevoflurane

SUMMARY:
This study compares desflurane with sevoflurane for school-age children in postoperative cognitive function.

DETAILED DESCRIPTION:
The postoperative cognitive dysfunction (POCD) of school-age children (6-14 age) after operation draw more attention from both society and family. It is well known that, compare with sevoflurane, desflurane could improve cognitive function in elderly patients. But whether Desflurane could improve postoperative cognitive function compare with Sevoflurane for the school-age children, there is no consistent conclusion.

ELIGIBILITY:
Inclusion Criteria:

* 6-14 age, elective no-cardiac and non-neurological surgery , ASA physical statusⅠorⅡ, no preoperative cognitive function impairment, cooperate to complete the entire test.

Exclusion Criteria:

* Allergic to halogens inhaled anesthetics, malignant hyperthermia susceptible patients, intracranial hypertension, emotional disorder, hyperactivity, history of operation, mental retardation, audio-visual obstacles, history of congenital heart disease, Important organ dysfunction, history of drug abuse
* History of epilepsy
* Preoperative respiratory infection significantly.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative cognitive dysfunction | Within 7 days after operation
  Cognitive function score should be carried out for all children at preoperative 1d, postoperative 2 d, 3d and 7d. If postoperative score compared with preoperative score drop 1 points or more, then postoperative cognitive dysfunction will be recorded.

SECONDARY OUTCOMES:
age | 1 day before operation
  years old
male | 1 day before operation
  If the child is boy,it's "yes",or it's "no".
height | 1 day before operation
  CM
weight | preoperation
  kg
previous operation history | preoperation
  If the child had previous operation history,it's "yes",or it's "no".
the duration of anesthesia | From the time began to give the anesthetic to the time of pull out the endotracheal intubation
  minutes
the duration of operation | Surgery end time minus the start time
  minutes
total blood loss | The total blood loss of the whole surgery time.
  ml
total volume of infusion | The total volume of infusion of the whole surgery time.
  ml
whether there is respiratory depression in postanesthesia care unit | The period which the patient stay at post anesthesia care unit,from the time enter to postanesthesia care unit to the time leave postanesthesia care unit,the estimated period is up to 30 minutes.
  If the child has respiratory depression during this time,it's "yes",or it's "no".
the length of hospital stay | the time from admission to hospital to discharge from hospital,the estimated period is up to 5 days.
  days
S100β | 1 day after surgery
  obtain the children's plasma to detection S100β with ELEASE.
NSE | 1 day after surgery
  obtain the children's plasma to detection NSE with ELEASE.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Radtke FM, Franck M, Herbig TS, Papkalla N, Kleinwaechter R, Kork F, Brockhaus WR, Wernecke KD, Spies CD. Incidence and risk factors for cognitive dysfunction in patients with severe systemic disease. J Int Med Res. 2012;40(2):612-20. doi: 10.1177/147323001204000223. PMID 22613422
- [Result] Bekker AY, Weeks EJ. Cognitive function after anaesthesia in the elderly. Best Pract Res Clin Anaesthesiol. 2003 Jun;17(2):259-72. doi: 10.1016/s1521-6896(03)00005-3. PMID 12817919
- [Result] Mckay RE, Large MJC, Balea MC, Mckay WR. Airway reflexes return more rapidly after desflurane anesthesia than after sevoflurane anesthesia. Anesth Analg. 2005 Mar;100(3):697-700. doi: 10.1213/01.ANE.0000146514.65070.AE. PMID 15728054
- [Result] Arslan M, Kurtipek O, Dogan AT, Unal Y, Kizil Y, Nurlu N, Kamaci S, Kavutcu M. Comparison of effects of anaesthesia with desflurane and enflurane on liver function. Singapore Med J. 2009 Jan;50(1):73-7. PMID 19224088
- [Result] Rortgen D, Kloos J, Fries M, Grottke O, Rex S, Rossaint R, Coburn M. Comparison of early cognitive function and recovery after desflurane or sevoflurane anaesthesia in the elderly: a double-blinded randomized controlled trial. Br J Anaesth. 2010 Feb;104(2):167-74. doi: 10.1093/bja/aep369. Epub 2009 Dec 30. PMID 20042477
- [Result] Locatelli BG, Ingelmo PM, Emre S, Meroni V, Minardi C, Frawley G, Benigni A, Di Marco S, Spotti A, Busi I, Sonzogni V. Emergence delirium in children: a comparison of sevoflurane and desflurane anesthesia using the Paediatric Anesthesia Emergence Delirium scale. Paediatr Anaesth. 2013 Apr;23(4):301-8. doi: 10.1111/pan.12038. Epub 2012 Oct 9. PMID 23043512
- [Result] Dexter F, Bayman EO, Epstein RH. Statistical modeling of average and variability of time to extubation for meta-analysis comparing desflurane to sevoflurane. Anesth Analg. 2010 Feb 1;110(2):570-80. doi: 10.1213/ANE.0b013e3181b5dcb7. Epub 2009 Oct 9. PMID 19820242
- [Result] Valley RD, Freid EB, Bailey AG, Kopp VJ, Georges LS, Fletcher J, Keifer A. Tracheal extubation of deeply anesthetized pediatric patients: a comparison of desflurane and sevoflurane. Anesth Analg. 2003 May;96(5):1320-1324. doi: 10.1213/01.ANE.0000058844.77403.16. PMID 12707126
- [Result] Tachibana S, Hayase T, Osuda M, Kazuma S, Yamakage M. Recovery of postoperative cognitive function in elderly patients after a long duration of desflurane anesthesia: a pilot study. J Anesth. 2015 Aug;29(4):627-30. doi: 10.1007/s00540-015-1979-y. Epub 2015 Feb 1. PMID 25638572